CLINICAL TRIAL: NCT02265926
Title: Respiratory Consequences of N95-type Mask Usage in Pregnant Healthcare Workers - A Controlled Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Pearl Tong, Associate Consultant, National University Health System, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/00226
Record Dates: First submitted 2014-09-13; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Hypoventilation
Keywords: filtering facepiece respirators; N95 masks; pandemic response; pregnant healthcare workers
MeSH Terms: conditions — Hypoventilation | interventions — N95 Respirators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N95 (Experimental): Intervention: N95 mask material
  Interventions: Device: N95 mask

INTERVENTIONS:
Device: N95 mask — N95 mask material used to cover aperture of Hans Rudolph mask

SUMMARY:
The study aims to find out if usage of N95 type respirators affects respiratory parameters in pregnant women so as to provide guidance on N95 respirator usage in pregnant healthcare workers.

DETAILED DESCRIPTION:
The first phase of the study aims to determine the average workload of a nurse. In the second phase of the study, this workload is then translated to walking on a treadmill while pregnant subjects wore special masks open to air, then occluded with N95 mask materials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had spontaneously conceived singleton pregnancies and were between 21 to 40 years old. Their hemoglobin levels were ≥11g/dL

Exclusion Criteria:

* Any cardiorespiratory illness, influenza-like illness in the week prior to the trial, or any pregnancy-related complications such as gestational diabetes, hypertension, intrauterine growth restriction, placenta previa, ruptured membranes, or threatened preterm labor. Any neuromuscular conditions that would preclude them from using the treadmill.

Haemoglobinopathies.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Minute Ventilation | 15 minutes
  Participants wore a tight fitting mask (Hans Rudolph) that was attached to the metabolic cart through an air sampling tube. Inspired ambient air and expired air were channeled through a pneumotachometer that was attached to the front of the mask which calculated air volume by the rate of rotation of a rotor turbine located within it. The turbine had zero resistance to air flow and the rate of rotation of the turbine, sensed by infrared light within the pneumotachometer, corresponds directly to inspired and expired air volume for each breath. Multiple air samples from each expired-breath was drawn into the metabolic carts through a sampling line for the measurement of oxygen and carbon dioxide content by the respective gas sensors within the metabolic carts.

SECONDARY OUTCOMES:
Oxygen and carbon dioxide exchanged | 15 minutes
  Participants wore a tight fitting mask (Hans Rudolph) that was attached to the metabolic cart through an air sampling tube. Inspired ambient air and expired air were channeled through a pneumotachometer that was attached to the front of the mask which calculated air volume by the rate of rotation of a rotor turbine located within it. The turbine had zero resistance to air flow and the rate of rotation of the turbine, sensed by infrared light within the pneumotachometer, corresponds directly to inspired and expired air volume for each breath. Multiple air samples from each expired-breath was drawn into the metabolic carts through a sampling line for the measurement of oxygen and carbon dioxide content by the respective gas sensors within the metabolic carts.

CONTACTS AND LOCATIONS:
Overall Officials: Eu-Leong Yong, PhD, Principal Investigator — NUHS
Locations (1):
- NUHS, Singapore, Singapore